CLINICAL TRIAL: NCT05421325
Title: Assessment of QBKPN Site-Specific Immunomodulator (SSI) Efficacy in Improving Innate Immune Function and Reducing All-Cause Respiratory Tract Infection Morbidity in Adults 65 Years of Age or Older Residing in the Community, in Independent-Living, Assisted-Living and Long-term Care Facilities
Brief Title: Efficacy of QBKPN Site-Specific Immunomodulator in Improving Innate Immune Function & Reducing Respiratory Tract Infection in Older Adults
Acronym: RESILIENCE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qu Biologics Inc. (Industry)
Collaborators: The National Research Council of Canada Industrial Research Assistance Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QBKPN-IS-01
Record Dates: First submitted 2022-05-11; First posted 2022-06-16 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Immune Deficiency
Keywords: Immunosenescence; immunodegeneration; immune dysfunction; older adult
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QBKPN SSI (Experimental): QBKPN SSI (0.1 mL) by subcutaneous injection 3 times per week (Monday, Wednesday & Friday) for 4 weeks.
  Interventions: Biological: QBKPN SSI
- Placebo (Placebo Comparator): Placebo (Normal Saline) (0.1 mL) by subcutaneous injection 3 times per week (Monday, Wednesday & Friday) for 4 weeks.
  Interventions: Other: Normal Saline Placebo

INTERVENTIONS:
Biological: QBKPN SSI — Site-Specific Immunomodulator
  Arms: QBKPN SSI
Other: Normal Saline Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
This study is designed to test whether QBKPN SSI can improve immune function in older adults, including how well it can protect against respiratory and other infections, whether it improves the body's response to COVID-19 vaccines, what effect it has on maintaining or improving quality of life, activity level and health status and whether it has an effect on glycemic control.

QBKPN is a new medication in a class known as Site-Specific Immunomodulators (SSI). SSIs are designed to train and/or improve innate immune function to reduce the risk of infections, improve immune response to cancer, and slow the progression of chronic inflammatory diseases.

It is believed that QBKPN SSI can work with the immune system to help protect against respiratory and other infections.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of adults 65 years of age or older residing in the community, in independent-living, assisted-living and long-term care (LTC) facilities to assess the effect of QBKPN SSI on improvement of innate immunity and reduction of all-cause respiratory tract infection morbidity.

Approximately 72 participants will be enrolled; approximately 36 from the community and independent-living facilities and approximately 36 from assisted-living and LTC facilities.

Eligible participants will be screened and enrolled by study staff, who will conduct all study visits, and administer or teach self-administration of study treatment. Blood/sample collections will be performed by study staff or by staff at Vancouver Coastal Health Research Institute Clinical Research Unit. Participants will have the options of nurse-administration, self-administration or a combination of nurse- and self-administration of study treatment. Participants will receive study treatment for 4 weeks then be monitored for 22 weeks. Blood/urine sampling will be performed at Baseline, Weeks 4, End of Treatment, Week 8, Week 12 and Week 26. A phone call visit will be conducted at Week 20.

Immunological testing for trained innate immunity, capacity for anti-viral innate immune response, measures of immune augmentation, duration of adaptive immune response to SARS-CoV-2 vaccination and/or infection, change in metabolome and Natural Killer (NK) cell function will be performed.

Safety and tolerability of study treatment will be assessed through clinical laboratory parameters and treatment-emergent adverse events.

Clinical benefits of study treatment will be assessed via medical record review and patient-reported outcomes. Study staff will record any confirmed/probable/possible infections (viral and bacterial, including respiratory and non-respiratory), any microbiologic or radiologic testing performed to investigate for infection, any prescribed antibiotics/antivirals and duration of treatment and reason for and duration of any hospitalizations.

Clinical assessments will also include frailty index (Rockwood Clinical Frailty Scale), quality of life [Dementia Quality of Life Questionnaire(DEMQOL)], end-of-life prediction score (CHESS Scale) and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Be a resident of the community or a long-term care, independent-living or assisted living facility participating in the study
2. Be aged 65 years or older
3. Be able to provide written, informed consent themselves
4. Male subjects engaged in vaginal intercourse with women of childbearing potential must be surgically sterile or agree to practice effective barrier contraception during the entire study treatment period (4 weeks) and one month after the last dose of study drug or agree to completely abstain from vaginal intercourse with women of childbearing potential during this period.

Exclusion Criteria:

1. Life expectancy of less than 3 months due to terminal illness as determined by the Study Investigator
2. Taking biologic immunosuppressive agents (e.g., Anti-Tumour Necrosis Factor Alpha (anti-TNFa) antibodies, rituximab, ibrutinib, imatinib) calcineurin inhibitors, myelosuppressants (e.g., methotrexate, mycophenolate), or other systemic immunosuppressants. Note: NSAIDs, colchicine, aspirin and oral glucocorticoids at a dose equivalent to less than or equal to 5mg prednisone per day are allowed
3. Currently being treated or less than 30 days from being treated for confirmed or probable infection with systemic (i.e., not topical) antibiotics or antivirals
4. Have a known allergy or hypersensitivity to killed whole-cell bacterial vaccines
5. Any condition that, in the opinion of the Investigator, would preclude the person from participation in the study due to safety or monitoring concerns
6. Any treatment with experimental or investigational therapies within 3 months prior to Screening and/or any planned treatment with experimental or investigational therapies during the entire course of study participation
7. On current treatment for active malignancies (e.g., chemotherapy, radiation) or planned cancer surgery during the study period. Note: People on exclusively hormonal therapy for breast or prostate cancer are allowed. People with prior or planned surgery for localized squamous cell or basal cell carcinoma of the skin are allowed

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate innate immune training in participants treated with QBKPN SSI compared to placebo. | Baseline to End of Treatment (EOT) (Week 4)
  Innate immune training will be measured by change in stimulated IL-β using RBM Myriad's TLR4 ligand (LPS) TruCulture Tube assay.
Incidence of treatment-emergent adverse events (safety & tolerability) in participants treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4) and Week 8
  Treatment-emergent adverse events assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Change in clinical laboratory parameters (safety & tolerability) measured by blood hematology analysis in participants treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4) and Week 8
  Hematology analysis includes: Hematocrit (Hct), Hemoglobin (Hgb), Mean Corpuscular Hemoglobin (MCH), Mean Corpuscular Hemoglobin Concentration (MCHC), Mean Corpuscular Volume (MCV), platelet count, Red Blood Cell (RBC) count, White Blood Cell (WBC) count with differential.
Change in clinical laboratory parameters (safety & tolerability) measured by blood chemistry analysis in participants treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4) and Week 8
  Clinical chemistry analysis includes: Alanine Aminotransferase (ALT), Albumin (ALB), Alkaline Phosphatase (ALK-P), Aspartate Aminotransferase (AST), bilirubin, Gamma-Glutamyl Transferase (GGT), creatinine, estimated Glomerular Filtration Rate (eGFR), C-Reactive Protein (CRP), electrolytes.
Change in clinical laboratory parameters (safety & tolerability) measured by urinalysis in participants treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4) and Week 8
  Urinalysis includes: blood, glucose, ketones, leukocyte esterase, nitrite, pH, protein and specific gravity.

SECONDARY OUTCOMES:
Evaluate capacity for anti-viral innate immune response by measuring change in stimulated type I and type III interferon production in participants treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4)
  Type I and type III interferon production measured using RBM Myriad's Toll-like Receptor 7/8 agonist (TLR7/8) (Resiquimod R848) TruCulture Tube assay.
Difference in incidence of all-cause respiratory tract infections assessed by medical record review in participants treated with QBKPN SSI compared to placebo. | Baseline to Week 26
  Respiratory tract infections identified using revised McGeer Criteria and/or as determined by participants' medical providers.
Difference in incidence of all-cause respiratory tract infections assessed by patient reported outcomes (PROs) in participants treated with QBKPN SSI compared to placebo. | Baseline to Week 26
  Respiratory tract infections identified using revised McGeer Criteria and/or as determined by participants' medical providers
Difference in severity of all-cause respiratory tract infections assessed by medical record review in participants treated with QBKPN SSI compared to placebo. | Baseline to Week 26
  Severity of all-cause respiratory tract infections measured using World Health Organization (WHO) 8-point ordinal scale for respiratory viral infections [minimum score 0 (uninfected) to maximum score 8 (death)] and Pneumonia Severity Index (PORT Score) (minimum: Class I, 0.1% mortality to maximum: Class V, 27% mortality) for respiratory bacterial infections. [Note: if source of infection is unknown, both WHO 8-point ordinal scale and PORT score will be collected.]
Difference in severity of all-cause respiratory tract infections assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Severity of all-cause respiratory tract infections measured using World Health Organization (WHO) 8-point ordinal scale for respiratory viral infections and Pneumonia Severity Index (PORT Score) for respiratory bacterial infections. [Note: if source of infection is unknown, both WHO 8-point ordinal scale and PORT score will be collected.]
Difference in symptom duration of all-cause respiratory tract infections assessed by medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Symptom duration assessed by medical record review
Difference in symptom duration of all-cause respiratory tract infections assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Symptom duration assessed by PROs
Number of courses of antibiotic/antiviral drugs prescribed for respiratory infections assessed by medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Number of courses of antibiotic/antiviral drugs assessed by medical record review
Number of courses of antibiotic/antiviral drugs prescribed for respiratory infections assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Number of courses of antibiotic/antiviral drugs assessed by PROs
Difference in incidence of all-cause non-respiratory infection assessed by medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  All-cause non-respiratory infection identified using revised McGeer Criteria and/or as determined by participants' medical providers
Difference in incidence of all-cause non-respiratory infection assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  All-cause non-respiratory infection identified using revised McGeer Criteria and/or as determined by participants' medical providers
Difference in severity of all-cause non-respiratory infection assessed by medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Severity of all-cause non-respiratory infection assessed by medical record review
Difference in severity of all-cause non-respiratory infection assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Severity of all-cause non-respiratory infection assessed by PROs
Difference in severity of all-cause non-respiratory infection assessed by hospitalizations due to non-respiratory infections in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Severity of all-cause non-respiratory infection assessed by hospitalizations due to non-respiratory infections
Difference in severity of all-cause non-respiratory infection assessed by mortality due to non-respiratory infections in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Severity of all-cause non-respiratory infection assessed by mortality due to non-respiratory infections
Difference in symptom duration of all-cause non-respiratory infection assessed via medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Symptom duration assessed via medical record review
Difference in symptom duration of all-cause non-respiratory infection assessed by PROs in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  Symptom duration assessed by PROs
Number of courses of antibiotic/antiviral drugs prescribed for non-respiratory infections assessed by medical record review in participants treated with QBKPN SSI compared to placebo | Baseline to Week 26
  assessed by medical record review
Number of courses of antibiotic/antiviral drugs prescribed for non-respiratory infections assessed by PROs in participants treated to QBKPN SSI compared to placebo | Baseline to Week 26
  Number of courses of antibiotic/antiviral drugs assessed by PROs
Change in quality of life as measured by Dementia Quality of Life (DEMQOL) Scale in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4) and Weeks 8, 12 & 26
  Quality of life measured using DEMQOL Scale. Scores are from 28 to 112; higher scores indicate better quality of life
Change in frailty as measured by the Rockwood Clinical Frailty Scale in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4) and Weeks 8, 12 & 26
  Frailty measured using Rockwood Clinical Frailty Scale. Scores are from minimum of 1 (very fit) to maximum of 7 (severely frail)
Change in end-of-life prediction score as measured by Changes in Health, End-Stage Disease and Signs and Symptoms (CHESS) scale in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4) and Weeks 8, 12 & 26
  End-of-life prediction score measuring using CHESS scale. Scores are from minimum 0 (no health instability) to 5 (very high health instability)
Change in all-cause mortality in participants treated with QBKPN SSI compared to placebo | Up to 26 weeks after first dose of study drug
  Recording all-cause mortality

OTHER OUTCOMES:
Change in additional measures of plasma immune biomarkers that regulate innate & adaptive immune function augmentation measured using TruCulture Tube® assay (under stimulated & unstimulated conditions) of 48 analytes (cytokines & chemokines) | Baseline to EOT (Week 4) and Weeks 8, 12 and 26
  Plasma immune biomarkers measured using TruCulture Tube assay (under stimulated and unstimulated conditions) of 48 analytes (cytokines & chemokines) using multiplex technology assessment
Evaluation of duration of adaptive immune response to SARS-CoV-2 vaccination and/or infection measured by change in Cluster of Differentiation 4+ (CD4+) and Cluster of Differentiation 8+ (CD8+) T-cell response to SARS-CoV-2 S protein-derived peptides | Baseline to EOT (Week 4) and Weeks 8, 12 and 26
  Adaptive immune response measured by CD4+ and CD8+ T-cell response to SARS-CoV-2 S protein-derived peptides
Evaluation of duration of adaptive immune response to SARS-CoV-2 vaccination and/or infection measured by change in SARS-CoV-2 anti-S antibody titer in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4) and Weeks 8, 12 and 26
  Adaptive immune response to SARS-CoV-2 vaccination and/or infection measured by SARS-CoV-2 anti-S antibody titer
Evaluation of duration of adaptive immune response to SARS-CoV-2 vaccination and/or infection measured by change in SARS-CoV-2 anti-S antibody secretion from antigen stimulated Peripheral Blood Mononuclear Cells (PBMCs) | Baseline to EOT (Week 4) and Weeks 8, 12 and 26
  Adaptive immune response to SARS-CoV-2 vaccination and/or infection measured by SARS-CoV-2 anti-S antibody secretion from antigen stimulated Peripheral Blood Mononuclear Cells (PBMCs) in participants treated with QBKPN versus placebo
Change in plasma metabolome measured using mass spectrometry (untargeted) to assess which metabolites are significantly changed by treatment and which may predict response to treatment in patients treated with QBKPN SSI compared to placebo. | Baseline to EOT (Week 4) and Weeks 8, 12 and 26
  Change in plasma metabolome measured using untargeted mass spectrometry
Assessment of correlation of Immunoglobulin G (IgG) antibodies to K.variicola with the NK cell function and innate immune training in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4) and Week 26
  Correlation assessed by quantification of IgG antibodies to K. variicola and correlation with NK Vue assay and RBM Myriad's TLR4 ligand (LPS) TruCulture Tube assay results
Evaluation of durability of QBKPN SSI beyond EOT in participants treated with QBKPN SSI compared to placebo | Up to 26 weeks after first dose of study drug
  Durability of QBKPN SSI assessed by measuring innate immune training (see Outcome #1), anti-viral innate immunity (see Outcome #6), circulating Natural Killer (NK) cell function (see Outcome #37), all-cause respiratory and non-respiratory infections (see Outcomes #7 to #24)
Assessment of glycemic control through hemoglobin A1C (HbA1c) in participants treated with QBKPN compared to placebo | Baseline to EOT (Week 4) and Weeks 8, 12 & 26.
  Change in HbA1c
Assessment of NK cell function in participants treated with QBKPN SSI compared to placebo | Baseline to EOT (Week 4)
  NK cell function assessed by measuring stimulated IFN-y production using the NK Vue assay

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Steiner, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Qu Biologics Trial Site, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No